CLINICAL TRIAL: NCT00050479
Title: Preliminary Multi-Center Assessment of Laser and Medical Treatment of Diabetic Macular Edema
Brief Title: Laser and Medical Treatment of Diabetic Macular Edema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030065; 03-EI-0065
Record Dates: First submitted 2002-12-09; First posted 2002-12-10 (Estimated); Last update posted 2006-07-19 (Estimated); Status verified 2006-07

CONDITIONS: Macular Degeneration
Keywords: Types 1 and 2 diabetes; Diode Laser Photocoagulation; Elevated Low-Density Lipoprotein (LDL-C) Cholesterol
MeSH Terms: conditions — Macular Degeneration | interventions — Celecoxib

INTERVENTIONS:
Drug: Celecoxib (Celebrex)

SUMMARY:
This study will compare the side effects of two laser treatments for diabetic macular edema, a common condition in patients with diabetes. In macular edema, blood vessels in the retina, a thin layer of tissue that lines the back of the eye become leaky and the retina swells. The macula, the center part of the retina that is responsible for fine vision may also swell, causing vision loss. Traditional laser treatment (argon blue or green or yellow) for macular swelling, or edema, causes scarring that can expand and possibly lead to more loss of vision. Studies with a different type of laser (diode) may be less damaging. The results of this study on side effects of the treatments will be used to design a larger study of effectiveness. This study will also examine whether celecoxib (Celebrex® (Registered Trademark)), an anti-arthritis drug that reduces inflammation and swelling, can reduce inflammation and swelling of the retina. Patients with elevated cholesterol levels will be invited to participate in a cholesterol reduction part of the study to compare normal-pace cholesterol reduction with accelerated reduction.

Patients 18 years of age and older with type 1 or type 2 diabetes and macular edema that requires laser treatment may be eligible for this study. Candidates will be screened with the following tests and procedures:

* Medical history: to review past medical conditions and treatments.
* Physical examination: to measure vital signs (pulse, blood pressure, temperature, breathing rate) and examine the head and neck, heart, lungs, abdomen, arms and legs.
* Eye examination: to assess visual acuity (eye chart test) and examine pupils, lens, retina, and eye movements. The pupils will be dilated with drops for this examination.
* Blood tests: to measure cholesterol, blood clotting time, hemoglobin A1C (a measure of diabetes control), and to evaluate liver and kidney function.
* Eye photography: to help evaluate the status of the retina and changes that may occur in the future. Special photographs of the inside of the eye are taken using a camera that flashes a bright light into the eye. From 2 to 20 pictures may be taken, depending on the eye condition.
* Fluorescein angiography: to evaluate the eye's blood vessels. A yellow dye is injected into an arm vein and travels to the blood vessels in the eyes. Pictures of the retina are taken using a camera that flashes a blue light into the eye. The pictures show if any dye has leaked from the vessels into the retina, indicating possible blood vessel abnormality.

Participants will be randomly assigned to take celecoxib or placebo (an inactive, look-alike pill). Participants who have elevated cholesterol levels may return for a brief visit after 1 month. All patients will return for follow-up visits at 3, 6, and 12 months. Patients who require laser treatment will be randomly assigned to one of the two laser treatments. For these procedures, eye drops are put in the eye to numb the surface and a contact lens is placed on the eye during the laser beam application. Several visits may be required for additional laser treatments. The maximum number of treatments depends on how well the treatment is working. Patients who respond well to the study medication may receive no laser treatments. After the first year, patients will be followed every 6 months until either the patient returns for a 3-year visit, the last enrolled patient returns for the 1-year visit, or the patient requests to leave the study. During the follow-up visits, patients' response to treatment will be evaluated with repeat tests of several of the screening exams.

DETAILED DESCRIPTION:
This randomized pilot study is an important first step in planning a large multi-center clinical trial to evaluate medical and laser approaches that could improve the visual outcome for patients with diabetic retinopathy. This study will provide preliminary safety data on these therapies as well as allow for assessment of the performance of ocular outcomes and study design for use in subsequent trials. If there are no safety concerns, the results of this pilot will be helpful in the design of a large multicenter clinical trial by providing data on estimates of expected treatment effects.

Using a factorial design, this study will compare (1) diode (micropulse) laser photocoagulation to mild ETDRS style focal photocoagulation and, (2) treatment with a COX-2 inhibitor (celecoxib), or placebo prior to and following laser photocoagulation. The primary outcomes are a visual acuity drop or increase of 15 letters or more from baseline to year 3. The secondary outcome is a significant reduction in macular edema, defined as a 50% reduction in thickening as measured by Optical Coherence Tomography (OCT), a two step reduction in macular thickness compared to standard stereoscopic fundus photographs, and a 50% reduction in the area of leakage as measured by fluorescein angiography. The University of Wisconsin Fundus Photography Reading Center will grade OCT, photographs, and angiograms and will be masked to treatment assignment. Other secondary outcomes will include the timing of the first required laser treatment, changes in visual acuity throughout the study, and the number of laser treatments required during the course of the study. In addition, all adverse events and abnormal laboratory values will be collected and tabulated. Specific objectives regarding safety and efficacy follow:

Safety

Is the risk of visual loss in patients with clinically significant diabetic macular edema potentially different across treatment groups?

Preliminary Assessment of Potential Outcomes

Is there evidence that any treatment combinations could be effective in reducing retinal thickening?

Is there evidence that celecoxib may inhibit or induce retinal thickening?

What are the estimated treatment effects on vision?

Is the number of laser treatments required to achieve a reduction in retinal thickening similar across treatment groups?

The tertiary objective of this study will be to examine the effects of dramatically reducing low-density lipoproteins cholesterol in patients with diabetic macular edema and elevated serum lipid levels. Change vision and retinal thickness will be compared across three groups; (1) patients without elevated serum lipids at baseline, (2) patients with elevated lipid levels at baseline and receive standard of care treatment, and (3) patients with elevated lipid levels at baseline and are aggressively treated pharmacologically.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for the study each participant must have at least one eye, which satisfies all ocular inclusion criteria:

1. Participants with type 1 or 2 diabetes.
2. Participants with clinically significant macular edema in at least one eye that requires laser treatment, but in the opinion of the Investigator, can be delayed for up to at least 3 months.
3. Best corrected visual acuity 20/400 or better as measured on an ETDRS chart in the eye with clinically significant macular edema; this eye will be considered they study eye. If both eyes have clinically significant macular edema and best corrected visual acuity greater than or equal to 20/400, the right eye will be considered the study eye, however, both eyes will be eligible for treatment.
4. May have had proliferative diabetic retinopathy but scatter photocoagulation must have been performed more than four months ago.
5. Ocular media sufficiently clear to allow for quality fundus photography.
6. If aphakic or pseudophakic, lens removal must have occurred at least 6 months prior to enrollment.
7. Documented hemoglobin A1C 12% or less within one month of baseline.
8. Willingness to accept randomization for diet or drug therapy for lowering of elevated lipid levels (for sites participating in the Lipid Lowering study option).
9. Understand and sign the informed consent.
10. Participants 18 years of age and older since the population of interest is primarily adults.

EXCLUSION CRITERIA:

To be eligible for the study, each participant must not satisfy an ocular exclusion cirterion in both eyes.

1. Retinopathy that requires scatter photocoagulation immediately.
2. Ocular disease other than diabetic retinopathy that may confound the outcome of the study (e.g. age-related macular degeneration, drug toxicity, uveitis, etc.).
3. Prior of current macular detachment in the eligible eye(s).
4. Use of an investigational drug within 30 days of enrollment.
5. Malaborsorption syndrome.
6. Concurrent administration of the anti-obesity drug orlistat (Xenical).
7. Positive serum pregnancy test or currently lactating for women of childbearing potential.
8. Chronic requirement (e.g., greater than or equal to 4 weeks at a time) for ocular medication for diseases that, in the judgement of the examining physician, are vision thereateniong or may affect the primary outcome (artificial tears are permitted).
9. History of cancer and prognosis of survival of less than 3 years.
10. Participants whose diabetic macular edema, in the opinion of the Principal Investigator, cannot benefit from laser treatments, including those with subretinal fibrosis, severe macular non-perfusion, or parafoveal leakage in oth eyes.
11. Participants that have a history of focal laser treatment, and in the opinion of the investigator are thought to be refractory (e.g., > 50 micron burns or equivalent) to laser treatment or wwere treated within 3 months of baseline.
12. Participants with clear vireal-retinal tracion wiich in the opinion of the investigator needs to be treated as a contributor macular edema.
13. Participants requiriing herapy with topaical ophthalmic prostaglandin analogues.
14. Laboratory values outside normal limits and considered clinically significant by the investigator.
15. Past or current liver disease, which precludes the use of the lipid-lowering drugs.
16. Used Celebrex [Registered Trademark] or any other COX-2 inhibitor, NSAIDs, or ocular topical NSAID use great than 3 days per week for a period of 4 weeks or more within 6 months prior to enrollment, or likely need during the study (Aspirin dose of 325 mg per day is permitted).
17. Concurrent warfarin therapy or known bleeding diathesis.
18. Concurrent lithium therapy.
19. History of peptic ulcer disease within 1 year prior to enrollment.
20. History of kidney disease (serum creatinine greater than 2.5 mg/dL, or need for dialysis).
21. Allergy to sulfa- containing compounds, NSAIDs, or demonstrtion of the aspirin triad.
22. History of inflammatory bowel disease.
23. History of mycardial infarction within 2 years prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2002-12; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Han DP, Mieler WF, Burton TC. Submacular fibrosis after photocoagulation for diabetic macular edema. Am J Ophthalmol. 1992 May 15;113(5):513-21. doi: 10.1016/s0002-9394(14)74722-1. PMID 1575225
- [Derived] Solomon SD, Wittes J, Finn PV, Fowler R, Viner J, Bertagnolli MM, Arber N, Levin B, Meinert CL, Martin B, Pater JL, Goss PE, Lance P, Obara S, Chew EY, Kim J, Arndt G, Hawk E; Cross Trial Safety Assessment Group. Cardiovascular risk of celecoxib in 6 randomized placebo-controlled trials: the cross trial safety analysis. Circulation. 2008 Apr 22;117(16):2104-13. doi: 10.1161/CIRCULATIONAHA.108.764530. Epub 2008 Mar 31. PMID 18378608